CLINICAL TRIAL: NCT07091097
Title: Multivisceral Oncological Resections Involving the Pancreas - An International Multicenter Study
Acronym: MORIP-AIMS
Status: Completed | Type: Observational
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Artur Rebelo, MD, Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: 2023-211
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer; Multivisceral Pancreatic Resections
Keywords: multivisceral resection, pancreatic malignancies, oncological resections, outcomes, risk factors.
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing multivisceral pancreatic resections: Concerning pancreatic malignancies, multivisceral pancreatic resection refers to the excision of organs beyond the pancreas or spleen in cases of distal pancreatectomy (DP). For multivisceral pancreaticoduodenectomies or total pancreatectomies, the resection encompasses additional organs other than the distal two-thirds of the stomach, duodenum with the first jejunal loop, bile duct including the gallbladder, and spleen. It is important to note that additional procedures like portal vein resection or splenectomy are not categorized as multivisceral resections within the respective resection types. In cases involving non-pancreatic malignancies, any surgical procedure that includes resection of the pancreas along with other organs will be classified as a multivisceral resection. Notably, patients who underwent isolated pancreatic resection for pancreatic metastasis or revision pancreatectomies will be excluded from this analysis. P

SUMMARY:
Background: Complete resection is the primary curative option for most non-metastatic solid malignancies. Locally advanced stages, involving adjacent organs or structures, may require multivisceral resection. This study aims to comprehensively assess outcomes and risk factors of multivisceral oncological resections involving the pancreas, enhance understanding, and provide clinical guidance. The potential establishment of an international study group, centered on multivisceral resections involving the pancreas, will be further pursued based on the insights derived from this study.

Objective: The objective of this study is to evaluate the outcomes of multivisceral oncological resections involving the pancreas and identify predictive factors for morbidity/mortality as well as for overall and disease-free survival.

Methods: This retrospective multicenter study involves centers on a global scale conducting multivisceral oncological resections involving the pancreas. Data will be collected retrospectively from January 1st, 2010 to December 31st, 2022. Eligible patients are those undergoing elective multivisceral oncological resections involving the pancreas. Patient and operation characteristics, perioperative therapies, outcomes, complications, resection margins, and survival are recorded. Statistical analysis includes appropriate tests and subgroup analyses for distinct tumor entities.

ELIGIBILITY:
Concerning pancreatic malignancies, multivisceral pancreatic resection refers to the excision of organs beyond the pancreas or spleen in cases of distal pancreatectomy (DP). For multivisceral pancreaticoduodenectomies or total pancreatectomies, the resection encompasses additional organs other than the distal two-thirds of the stomach, duodenum with the first jejunal loop, bile duct including the gallbladder, and spleen. It is important to note that additional procedures like portal vein resection or splenectomy are not categorized as multivisceral resections within the respective resection types. In cases involving non-pancreatic malignancies, any surgical procedure that includes resection of the pancreas along with other organs will be classified as a multivisceral resection. Notably, patients who underwent isolated pancreatic resection for pancreatic metastasis or revision pancreatectomies will be excluded from this analysis. Patients who were not undergoing oncological resections (e. g. traumatic lesions) or those who did not undergo surgery as "curative intent" will be also excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Concerning pancreatic malignancies, multivisceral pancreatic resection refers to the excision of organs beyond the pancreas or spleen in cases of distal pancreatectomy (DP). For multivisceral pancreaticoduodenectomies or total pancreatectomies, the resection encompasses additional organs other than the distal two-thirds of the stomach, duodenum with the first jejunal loop, bile duct including the gallbladder, and spleen. It is important to note that additional procedures like portal vein resection or splenectomy are not categorized as multivisceral resections within the respective resection types. In cases involving non-pancreatic malignancies, any surgical procedure that includes resection of the pancreas along with other organs will be classified as a multivisceral resection. Notably, patients who underwent isolated pancreatic resection for pancreatic metastasis or revision pancreatectomies will be excluded from this analysis. Patients who were not undergoing oncological resections (
Sampling Method: Non-Probability Sample
Enrollment: 1283 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Mortality | 90 Day
  Mortality after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Uniklinikum Halle, Halle, Germany

IPD SHARING:
Plan to Share IPD: Undecided